CLINICAL TRIAL: NCT04317482
Title: The Human Stress Response in a Simulated ED Setting
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 260721
Record Dates: First submitted 2020-03-16; First posted 2020-03-23 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Stress Physiology; Stress Reaction; Substance Use Disorders; Methamphetamine-dependence; Stress, Emotional
Keywords: Stress Response
MeSH Terms: conditions — Fractures, Stress; Substance-Related Disorders; Stress, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard social stress task (Other): Participants will be given 4.5 minutes to prepare a 4.5-minute public speech on three standard scenarios presented in counterbalanced order. This will involve approximately 30 minutes of public speaking stress given expected transitions. The public speeches will be presented in front of 1-2 individuals who are evaluating their presentations. Immediately after the public speaking task, participants will be asked to complete a mental arithmetic task for 15 minutes.
  Interventions: Behavioral: Standard social stress task
- Stressful experience in the ED (Other): Participants will be given 4.5 minutes to prepare a 4.5-minute public speech on three experiences surrounding their most stressful ED visit. These experiences are presented in counterbalanced order. This will involve approximately 30 of public speaking stress given expected transitions. The public speeches will be presented in front of 1-2 individuals who are evaluating their presentations. Immediately after the public speaking task, participants will be asked to complete a mental arithmetic task for 15 minutes.
  Interventions: Behavioral: Stressful experience in the ED

INTERVENTIONS:
Behavioral: Standard social stress task — Participants will be asked to respond in detail to three scenarios. This is a standard social stressor task. Participants may be prompted by an experimenter. However, the participant will receive no verbal nor nonverbal feedback.
  Arms: Standard social stress task
Behavioral: Stressful experience in the ED — Participants will be asked to imagine and then describe both feelings and bodily sensations experienced at their most stressful ED visit, in order to help them more fully re-experience the situation. In this regard, the second condition is more similar to stress imagery employed by Sinha et al, which elevated cortisol to a greater degree than a social stressor task. Participants may be prompted by an experimenter. However, the participant will receive no verbal nor nonverbal feedback.
  Arms: Stressful experience in the ED

SUMMARY:
Stress is important for health. As emergency departments (EDs) are often stressful places, a better understanding of the human stress response is important for understanding how and why patients respond as they do when they come to the ED. Since the investigators cannot take up space in the ED for research, the investigators will instead recruit 20 methamphetamine-using participants who are not currently in treatment and 10 healthy adult matched participants to a simulated ED room in the University of Arkansas for Medical Sciences (UAMS) Simulation Center. The investigators will have participants perform a stressor task involving public speaking and a simple arithmetic task. The investigators will see if this experiment can be made to be like being in an actual ED by varying what participants speak about in the task. By doing this, the investigators hope to find out several important things: 1) Is a stressor task feasible and acceptable to participants? 2) What does the stress response -- as measured by cortisol and alpha-amylase -- look like in these participants? 3) Does varying what participants talk about make the experiment seem more like an actual ED? 4) Do participants under stress show even mild symptoms of agitation as measured by clinical scales? If so, how often?

DETAILED DESCRIPTION:
Aim 1: Determine the feasibility and acceptability of an ED-relevant stressor task as compared to a standard social stressor task. The investigators hypothesize that an ED-relevant stressor task will be feasible, as measured by the ability to recruit/randomize/retain participants, and as acceptable to participants as a standard social stressor task.

Aim 2: Measure the stress response (alpha-amylase, cortisol, vital signs) in participants who undergo an ED-relevant stress task compared to a standard social stress task. The investigators hypothesize that norepinephrine release will be adequately assessed by salivary alpha-amylase and that an ED-relevant stressor task will elicit similar or greater physiological responses as a standard social stress task.

Aim 3: Evaluate the ED-representativeness of an ED-relevant stressor task compared to a standard social stressor task. Although both tasks will be performed in a simulated ED room in the UAMS Simulation Center, the investigators hypothesize that an ED-relevant task will be rated as more representative of an actual ED visit.

Aim 4: Evaluate ethological ratings of non-verbal behavior thought to indicate assertion and ratings of agitation using rating scales commonly employed in the clinical environment for this purpose. Participants undergoing stress sometimes display symptoms of assertion or agitation, but it is unknown when or how often this occurs. The investigators hypothesize that ethological ratings will be correlated with agitation scale scores and physiological changes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult
* 21-55 years of age
* Self-reported recent history of meth use that meets DSM-5 criteria for current meth use disorder
* Have been previously inside an ED as either a patient or visitor
* Able to construct a stressful mental script of ED experiences
* Body mass index (BMI) < 30
* Ability to read and understand English
* If matched control, no lifetime history of any recreational or non-prescribed drug use.

Exclusion Criteria:

* Eating/drinking/taking drugs or alcohol the morning before the experiment
* If smoker, not smoking the morning before the experiment
* Subjective or objective signs of intoxication or withdrawal from any substance
* History of any serious medical condition such as cardiovascular, endocrine, neurologic (seizures), or hepatic disease
* Pregnancy
* History of any mental illness
* Hypertensive (>150/90) or abnormal EKG at screening
* Use of any daily medication
* Any recent night shift work in the last 4 weeks
* Any travel across time zones in the last 14 weeks
* Participation in a similar study in the past year
* Refusal to allow videotaping

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-08-26 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Determine the feasibility and acceptability of an ED-relevant stressor task as compared to a standard social stressor task. | Up to 12 hours
  Measure feasibility and acceptability in the following ways: participant recruitment; the number of participants completing the experiment; and the acceptability ratings of the task after completion. The 9-point acceptability responses will be analyzed by calculating the mean and 95% confidence intervals for each question, then calculating a chi-square goodness of fit test across the 3 ranges of the scores.
  Answers to open-ended questions about participant experiences will be coded using conventional content analysis, as per Hsieh and Shannon. In this analysis, two research associates separately read through all the participants' qualitative responses and highlight key words which reflect the overall idea of the patient's response. After multiple reviews, 3-5 main categories will be identified which reflect responses of a similar nature. After categorization, a third research associate will make final decisions on the placement of individual responses.
Measure the stress response (alpha-amylase) in participants who undergo an ED-relevant stress task compared to a standard social stress task. | Up to 12 hours
  Compare alpha-amylase in participants randomized to a standard stressor task (i.e., with three standard scenarios) versus an ED-relevant stressor task (i.e., with stressful imagery).
Measure the stress response (cortisol) in participants who undergo an ED-relevant stress task compared to a standard social stress task. | Up to 12 hours
  Compare cortisol levels in participants randomized to a standard stressor task (i.e., with three standard scenarios) versus an ED-relevant stressor task (i.e., with stressful imagery).
Measure the stress response (systolic blood pressure) in participants who undergo an ED-relevant stress task compared to a standard social stress task. | Up to 12 hours
  Compare systolic blood pressure in participants randomized to a standard stressor task (i.e., with three standard scenarios) versus an ED-relevant stressor task (i.e., with stressful imagery).
Measure the stress response (diastolic blood pressure) in participants who undergo an ED-relevant stress task compared to a standard social stress task. | Up to 12 hours
  Compare diastolic blood pressure in participants randomized to a standard stressor task (i.e., with three standard scenarios) versus an ED-relevant stressor task (i.e., with stressful imagery).
Measure the stress response (heart rate) in participants who undergo an ED-relevant stress task compared to a standard social stress task. | Up to 12 hours
  Compare heart rate in participants randomized to a standard stressor task (i.e., with three standard scenarios) versus an ED-relevant stressor task (i.e., with stressful imagery).
Evaluate the ED-representativeness of an ED-relevant stressor task compared to a standard social stressor task. | Up to 12 hours
  Measure ED-representativeness in the following way: the ED-representativeness ratings of the task after completion. Investigators will compare representative ratings on a 9-point scale. The 9-point acceptability responses will be analyzed by calculating the mean and 95% confidence intervals for each question, then calculating a chi-square goodness of fit test.
Measure agitation scale ratings (Behavioral Activity Rating Scale) in participants who undergo an ED-relevant stress task compared to a standard social stress task. | Up to 12 hours
  Use the videotaped recordings to compare agitation scale ratings (Behavioral Activity Rating Scale) in participants randomized to a standard stressor task (i.e., with three standard scenarios) versus an ED-relevant stressor task (i.e., with three stressful ED experiences). Agitation will be rated on a 7-point scale (from "1 - difficult or unable to rouse" to "7 - violent, requires restraint").
Measure agitation scale ratings (Positive and Negative Syndrome Scale - Excited Component) in participants who undergo an ED-relevant stress task compared to a standard social stress task. | Up to 12 hours
  Use the videotaped recordings to compare agitation scale ratings (Positive and Negative Syndrome Scale - Excited Component) in participants randomized to a standard stressor task (i.e., with three standard scenarios) versus an ED-relevant stressor task (i.e., with three stressful ED experiences). Agitation will be rated on a 7-point scale (from "1 - absent" to "7 - extreme") on each of five items: poor impulse control, tension, hostility, uncooperativeness, and excitement.
Evaluate ethological ratings of non-verbal behaviors thought to indicate assertion using a rating scale (Ethological Coding System for Interviews) commonly employed in the clinical environment for this purpose. | Up to 12 hours
  Divide the videotaped recordings of the task into 15-second intervals and code for the presence or absence of non-verbal behaviors. These behaviors will then be calculated as a percentage (i.e., the number of time intervals with a behavior divided by the total number of time intervals). These will be compared participants randomized to a standard stressor task (i.e., with three standard scenarios) versus an ED-relevant stressor task (i.e., with three stressful ED experiences).

CONTACTS AND LOCATIONS:
Overall Officials: Alison Oliveto, Ph.D., Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No